CLINICAL TRIAL: NCT06332911
Title: International Multi-center Study to Confirm the Safety and Performance of the Shockwave™Peripheral Intravascular Lithotripsy Balloon for Advanced Endovascular Aortic Repair
Brief Title: Shockwave™Peripheral Intravascular Lithotripsy Balloon for Advanced Endovascular Aortic Repair
Acronym: TEVAR
Status: Recruiting | Type: Observational
Sponsor: Rede Optimus Hospitalar SA (Network)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RO-231129
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Thoracoabdominal Aortic Aneurysm, Without Mention of Rupture; Abdominal Aortic Aneurysm Without Rupture; Thoracic Aortic Aneurysm Without Rupture
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- complex endovascular thoracic aortic repair: Patients submitted to complex endovascular thoracic aortic repair with hostile iliac access vessels using the Shockwave device to gain access.
  Interventions: Device: Shockwave™ Peripheral Intravascular Lithotripsy Balloon M5+

INTERVENTIONS:
Device: Shockwave™ Peripheral Intravascular Lithotripsy Balloon M5+ — Cracking-not-debulking technique (SHOCKWAVE IVL)

SUMMARY:
Shockwave TEVAR is a nonrandomized, prospective, international, multi-center, PMCF, obervational study.

The aim of this study is to evaluate the outcomes of the Shockwave™ Peripheral Intravascular Lithotripsy Balloon (Shockwave Medical Inc.) in the routine treatment of hostile iliac accesses during TEVAR and F/BEVAR.

DETAILED DESCRIPTION:
Standardized forms will collect data on the performed procedure, underlying pathology, cardiovascular risks and information on preoperative examinations. Physiological parameters routinely measured prior, during and after any surgical intervention will be recorded as well. A 1 month, 6-months and 12-months follow-up visit will be conducted to assess adverse events and outcome of the index procedure.

In addition, this study aims to analyze the technical and procedure success to gain access via hostile iliac access vessels withShockwave Peripheral Intravascular Lithotripsy Balloon in patients submitted for complex endovascualre thoracic, throaco-abdominal or abdominal aortic repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (m/f) age ≥ 18 years at time of enrollment.
2. Diagnosis of thoracic and/or thoraco-abdominal (Extent I-V) and juxta/para-renal/short-neck aneurysm requiring the implantation of a thoracic and/or thoraco-abdominal fenestrated/branched aortic endograft with delivery system introducer sheath diameter equal or larger than 18 Fr (6 mm).
3. Hostile iliac access was defined in the presence of:

   * Heavily circumferential calcified iliac arteries
   * Inner diameter ≤ 6 mm
   * Severe stenosis (> 50%; > 2.5 m/s peak velocity; absence of triphasic duplex signal in ipsilateral common femoral artery)
4. We will accept the following presentations of aneurysm:

   * urgent cases,
   * elective,
   * symptomatic
   * and fast growing.
5. The repair was performed using Shockwave™ before the introduction of the main endograft. The iliac procedures can be accompanied by angioplasty and/or stent and stent-graft positioning.

Exclusion Criteria:

1. Patients submitted to surgical conduit bypass.
2. Not-severely calcified disease (absence of calcification).
3. In-stent restenosis/occlusion.
4. Inability to cross with 0.014 guidewire.
5. Any significant medical condition which, in the investigator's opinion, may interfere with the subject's optimal participation in the study.
6. Pre-stented iliac access vessels at the level of Shockwave implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient (m/f) age ≥ 18 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Technical success - defined as intention-to-treat basis | 30 days
  * Successful dilatation of the access vessels to 8mm without rupture
  * Successful endovascular access and deployment of all aortic devices
  * Performance of the Shockwave™ IVL: Includes the definition for technical success as well as delivery of the intended main endograft without the need for surgical conversion, arterial rupture and iliac artery occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, Dr., Study Director — Rede Optimus Hospitalar AG; Nikolaos Tsilimparis, Prof., Principal Investigator — Department of Vascular Surgery, LMU Hospital Munich
Locations (5):
- Germany (2):
  - Department of Vascular Surgery, LMU Hospital Munich, Münich, Bavaria
  - Department of Vascular Surgery, Klinikum Nürnberg Campus Süd, Nuremberg, Bavaria
- Italy (2):
  - University of Genoa School of Medicine, Ospedale Policlinico San Martino - HSM, Genoa, Liguria
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Veneto
- Inselspital, University Hospital Bern, Heart Vascular Center, Bern, Canton Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No